CLINICAL TRIAL: NCT01097265
Title: The Influence of Micrometastases on Prognosis and Survival in Stage I-II Colon Cancer Patients: The EnRoute+ Study
Brief Title: Study of Micrometastases in Patients With Stage I or Stage II Localized Colon Cancer That Can Be Removed by Surgery
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jeroen Bosch Ziekenhuis (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Diagnostic
Other Study IDs: JBZ-EnRoute+; CDR0000668525 (Registry Identifier: PDQ (Physician Data Query)); EUDRACT-2010-018612-32; EU-21016
Record Dates: First submitted 2010-03-31; First posted 2010-04-01 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2011-09

CONDITIONS: Colorectal Cancer
Keywords: stage I colon cancer; stage II colon cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — Capecitabine; Oxaliplatin; Watchful Waiting; Chemotherapy, Adjuvant; Sentinel Lymph Node Biopsy

INTERVENTIONS:
Drug: capecitabine
Drug: oxaliplatin
Other: active surveillance
Other: laboratory biomarker analysis
Procedure: adjuvant therapy
Procedure: lymph node mapping
Procedure: sentinel lymph node biopsy

SUMMARY:
RATIONALE: Diagnostic procedures such as sentinel lymph node mapping may help doctors find patients who are at risk of developing micrometastases and plan better treatment.

PURPOSE: This randomized phase II/III trial is studying micrometastases in patients with stage I or stage II localized colon cancer that can be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the subset of patients with stage I or II localized, resectable colon cancer (pN0) at risk for developing systemic metastases.
* To determine the clinical and prognostic relevance of occult nodal isolated tumor cells and micrometastases in these patients.
* To determine the benefits of adjuvant chemotherapy in patients with pN0micro+ colon cancer.

OUTLINE: This is a phase II feasibility study (stage 1) followed by a phase III multicenter, open-label, randomized, and controlled study (stage 2).

* Stage 1 (phase II feasibility study) After undergoing planned curative resection followed by ex vivo sentinel lymph node mapping (SLNM). Resected samples are examined. The sentinel lymph nodes of those deemed pN0 disease (no macroscopic metastases or angioinvasion) are further evaluated for micrometastases by serial sectioning and immunohistochemistry using pan-cytokeratin. pN0micro+ disease are defined as isolated tumor cells (ITC) < 0.2 mm or micrometastasis 0.2 - 2 mm. Patients with pN0 disease are followed-up once every 6 months for 3 years and then annually for 2 years.
* stage 2 (phase III randomized study): Patients undergo planned surgery and ex vivo SLNM as in stage 1. Patients with pN0micro- disease are assigned to arm C; patients with pN0micro+ disease are randomized to 1 of 2 intervention arms (arms A and B). .

  * Arm A (pN0micro+): Patients receive oral capecitabine twice daily on days 1-14 and oxaliplatin IV over 2 hours on day 1 OR oral capecitabine twice daily on days 1-14 alone according to standard protocol. Treatment repeats every 4 weeks for up to 8 courses. Patients are followed-up once every 6 months for 3 years and then annually for 2 years.
  * Arm B (pN0micro+): Patients are followed-up once every 6 months for 3 years and then annually for 2 years.
  * Arm C (pN0micro-): Patients are followed-up once every 6 months for 3 years and then annually for 2 years.
* .

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or radiologically confirmed primary colon cancer

  * Stage I or II disease
* Clinically localized disease judged potentially resectable for cure, without intraoperatively gross nodal involvement
* Planning to undergo elective resection of the tumor
* No histologically or radiologically confirmed locoregional lymph node or distant metastasis
* No disseminated disease
* No clinical tumor perforation or obstruction
* Patients enrolled in stage 2 and undergoing randomization must also meet the following criteria:

  * pN0micro+ disease as evidenced by detection of sentinel lymph node isolated tumor cells (<0.2 mm) or micrometastasis (0.2 - 2 mm)
  * No high-risk pN0 disease meeting any of the following criteria:

    * Less then 10 lymph nodes detected in resected specimen
    * Invasion in other organs (T4, Nx, Mx)
    * Colon perforation at presentation
    * Obstruction at presentation
    * Angioinvasion at pathological examination
  * No rectal cancer
  * No clinically positive nodal tumors or advanced disease (stage III or Dukes stage C disease)

PATIENT CHARACTERISTICS:

* Patients enrolled in stage 2 and undergoing randomization must also meet the following criteria:

  * WHO performance status 0-1 or American Society of Anesthesiologists Physical Status classification 1-2
  * Not pregnant or nursing
  * Able to comply with requirements of the study
  * Must be fit to undergo chemotherapy treatment
  * No other current serious illness or medical conditions, including any of the following:

    * Severe cardiac illness (NYHA class III-IV disease)
    * Significant neurologic or psychiatric disorders
    * Uncontrolled infections
    * Active disseminated intravascular coagulation
    * Other serious underlying medical conditions that could impair the ability of the patient to participate in the study
  * No known hypersensitivity to study drugs
  * No definite contraindications for the use of corticosteroids

PRIOR CONCURRENT THERAPY:

* No prior colorectal surgery
* Patients enrolled in stage 2 and undergoing randomization must also meet the following criteria:

  * No prior chemotherapy (for patients enrolled in stage 2 and undergoing randomization only)
  * At least 4 weeks since prior and no other concurrent experimental drugs
  * No concurrent immunosuppressive or antiviral drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2010-07; Primary Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Accrual rate (total number of pN0 patients included in the registration study monthly/center) (stage 1)
Rate of upstaging in pN0 colon cancer patients (stage 1)
Disease-free survival (DFS) at 3 years (stage 2)
Percentage of successful sentinel lymph node mapping procedures using multivariate analysis (stage 2)

SECONDARY OUTCOMES:
Overall survival (OS) at 3 years (stage 2)
Stratified analysis of DFS and OS according to total harvested lymph nodes per resected specimen and chemotherapy regimen (capecitabine and oxaliplatin versus capecitabine alone) (stage 2)

CONTACTS AND LOCATIONS:
Overall Officials: Koop Bosscha, MD, Principal Investigator — Jeroen Bosch Ziekenhuis
Locations (11):
- Netherlands (11):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Vrije Universiteit Medisch Centrum, Amsterdam
  - Netherlands Cancer Institute - Antoni van Leeuwenhoek Hospital, Amsterdam
  - Academisch Medisch Centrum at University of Amsterdam, Amsterdam
  - Catharina Ziekenhuis, Eindhoven
  - University Medical Center Groningen, Groningen
  - Leiden University Medical Center, Leiden
  - Academisch Ziekenhuis Maastricht, Maastricht
  - Universitair Medisch Centrum St. Radboud - Nijmegen, Nijmegen
  - University Medical Center Rotterdam at Erasmus Medical Center, Rotterdam
  - University Medical Center Utrecht, Utrecht

REFERENCES:
- [Result] Lips DJ, Koebrugge B, Liefers GJ, van de Linden JC, Smit VT, Pruijt HF, Putter H, van de Velde CJ, Bosscha K. The influence of micrometastases on prognosis and survival in stage I-II colon cancer patients: the Enroute plus sign in circle Study. BMC Surg. 2011 May 11;11:11. doi: 10.1186/1471-2482-11-11. PMID 21569373